CLINICAL TRIAL: NCT06035991
Title: Première Evaluation Clinique de la Transplantation Cardiaque de Greffons préservés à l'Aide d'un Système de Perfusion Ex-vivo prolongée
Brief Title: First Clinical Evaluation of Heart Transplantation With Grafts Preserved Using an Ex-vivo Extended Perfusion System
Acronym: PEGASE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ICAN Nutrition Education and Research (Industry); Centre Hospitalier Universitaire de la Guadeloupe (Other); University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP220091
Record Dates: First submitted 2023-07-24; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-07

CONDITIONS: Heart Transplantation
Keywords: Heart transplantation; XVIVO perfusion
MeSH Terms: interventions — Heart Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with end-stage Heart Failure (Experimental)
  Interventions: Procedure: Heart transplantation

INTERVENTIONS:
Procedure: Heart transplantation — Heart transplantation in patients who have obtained a favourable and motivated opinion from the Multidisciplinary Consultation Meeting (RCP) of the cardiac surgery department of the Hospital Pitié-Salpêtrière

SUMMARY:
The main objective of PEGASE is to validate the recovery of a satisfactory cardiac function of a transplanted heart after a prolonged period of preservation by an ex-vivo perfusion device. This recovery of cardiac function will have to happen within 15 days after transplantation.

DETAILED DESCRIPTION:
Heart transplantation is a scarce resource, only 1 patient among 2 had the opportunity to be grafted in France in 2022. Despite the shortage of organs, some potential heart transplants are currently not recovered because the ischemia duration anticipated before being grafted (from donor to recipient) is too long and not compatible with transplantation, actually limited to 4h, max.

Innovation in ex-vivo hypothermic perfusion allows to consider the extension of the graft viability time, thus offering the possibility of extending the pool of heart grafts available to the patients, The study aims to demonstrate the feasibility of taking heart grafts from donors in Martinique and Guadeloupe, transferring them via air transport and then successfully transplanting them to patients hospitalized in France, up to 14 hours later, using an ex-vivo cold perfusion device to protect the heart during transport.

Patients involved in this study will be patients in desperate need of transplantation, with no chance of receiving it, due to the French transplant allocation policy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients suffering from irreversible terminal heart failure with a medical indication for heart transplantation but who cannot be transplanted (per the graft allocation policy in France) or assisted (technical impossibility, contraindication, patient's refusal) and for whom a favourable and motivated opinion from the Multidisciplinary Consultation Meeting (RCP) of the cardiac surgery department of the Hospital Pitié-Salpêtrière has been made
* Having given their informed consent in writing

Exclusion Criteria:

* Technical obstacles which would generate an excessive surgical risk for the patient according to the medical opinion such as comorbidities or associated pathology not compatible with a transplant
* Known ongoing sepsis, defined as positive blood culture immediately prior to transplant (including with ventricular assist device)
* Candidate patient for Combined Organ Transplantation
* Patient protected by law (guardianship, curatorship, deprived of liberty)
* No affiliated with or entitled to a French social security scheme (AME included)
* Pregnant or breast-feeding female
* Current participation in another interventional study (category 1 of French Jardé law) or being in the exclusion period at the end of a previous study
* Patient unable to understand the information provided during the informed consent procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Short term recovery of Cardiac function | Within 15 days after transplantation
  Cardiac index greater than 2.5 L/min/m2 without inotropic support and/or temporary circulatory assistance (ECMO, IMPELLA, BCPIA) measured by thermodilution (SWAN-GANZ catheter) or echocardiography

SECONDARY OUTCOMES:
Survival | 15 days, 30 days, 9 months, 6 months and 12 months
Absence of cardiac deaths | 15 days, 30 days, 3 months, 6 months and 12 months
  Patient who survived or died for a reason other than failure of cardiac function
Cardiac function recovery | 30 days, 3months, 6 months and 12 months
  Cardiac index greater than 2.5 L/min/m2 without inotropic support and/or temporary circulatory assistance (ECMO, IMPELLA, BCPIA) measured by thermodilution (SWAN-GANZ catheter) or echocardiography
Adverse events after transplant | 15 days and 12 months
  * moderate or severe primary graft dysfunction (according to ISHLT consensus),
  * acute cell rejection >2R, VAD >1,
  * long-term circulatory support (LVAD, BiVAD, TAH)
Myocardial preservation | during the procedure/surgery
  Absence of significant edema (pre- and post-preservation graft weight)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEBRETON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data regulatory authority (CNIL, Commission Nationale de l'Informatique et des Libertés) do not allow for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal